CLINICAL TRIAL: NCT03066908
Title: A Prospective, Single Arm, Multicenter Study of the Sinopsys® Lacrimal Stent Used for Transcaruncular-Ethmoid Sinus Access and Saline Irrigation in Patients With Moderate to Severe Chronic Rhinosinusitis
Brief Title: Sinopsys Lacrimal Stent Study for Patients With Chronic Sinusitis or CRS
Acronym: CRS
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in study design
Sponsor: Sinopsys Surgical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLSUS05
Record Dates: First submitted 2017-02-17; First posted 2017-03-01 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Chronic Sinus Infection
Keywords: Chronic Rhinosinusitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Single Arm (Experimental): Sinopsys® Lacrimal Stent
  Interventions: Device: Sinopsys® Lacrimal Stent

INTERVENTIONS:
Device: Sinopsys® Lacrimal Stent — Transcaruncular paranasal sinus or nasal cavity access for the purpose of irrigating the ethmoid sinus with saline
  Other Names: SLS

SUMMARY:
A prospective, single arm, multicenter study designed to demonstrate that the Sinopsys® Lacrimal Stent can safely create transcaruncular access to the ethmoid sinus to enable sinus irrigation and reduce symptoms in patients with moderate to severe chronic rhinosinusitis.

ELIGIBILITY:
Inclusion Criteria:

* The Investigator has determined that the potential study subject has moderate to severe chronic rhinosinusitis with ethmoid involvement:
* Non-Contrast CT scan (coronal view) Total Zinreich Modified CT score of 10-41
* Inflammation/ involvement of the ethmoid sinus with left and/or right anterior ethmoid and/or posterior ethmoid Zinreich Modified CT scores of 1-4
* SNOT-22 total raw score ≥ 45
* Meets the American Academy of Otolaryngology - Head and Neck Surgery (AAO-HNS) criteria for chronic rhinosinusitis (CRS) (Rosenfeld, et al., 2007): 90 days or longer of two or more of the following signs and symptoms: Mucopurulent drainage (anterior, posterior, or both) Nasal obstruction (congestion) Facial pain-pressure-fullness, or Decreased sense of smell AND inflammation is documented by one or more of the following findings: Purulent (not clear) mucus or edema in the middle meatus or ethmoid region Polyps in nasal cavity or the middle meatus, and/or Radiographic imaging showing inﬂammation of the paranasal sinuses
* Has failed medical therapy (Rudmik, et al., 2016) defined as the following:

During the 90 days prior to enrollment, at a minimum:

One course of broad spectrum or culture directed oral antibiotic of at least 2 weeks duration 60 days of topical intranasal steroid therapy and; 30 days of saline irrigation

* Age ≥ 22 years
* Non-Contrast CT scan (coronal view) confirms depth of olfactory fossa is Keros classification type 1 or 2
* The potential study subject is capable of understanding and executing written informed consent (IC) and questionnaires/diaries in English

Exclusion Criteria:

* Sinus opacification score of <10 or > 41 measured using the Zinreich Modified CT scoring system
* Isolated sinus disease evident on Non-Contrast CT scan that would be unlikely to respond to target ethmoid treatment (e.g., isolated sphenoid, maxillary or frontal disease)
* Polyposis scored as 2 using the Modified Lund-Kennedy Score
* Prior ocular and/or sinus surgery that alter the boney anatomy or violate/enter the orbit or sinus in a way that would render these structures "non-intact" (i.e. FESS). Minor procedures such as balloon sinus dilation (>30 days), septoplasty or turbinectomy are not exclusions.
* Non-Contrast CT scan (coronal view) shows depth of olfactory fossa is Keros classification type 3
* Prior surgical history, physical exam, nasal endoscopy and/or imaging studies that suggest significant craniofacial deformity (such as any facial anatomic abnormality from surgical intervention, trauma, and congenital or any other cause thus prohibiting adequate placement of the Sinopsys Lacrimal Stent
* Presence of a sinonasal encepholocele as determined by Non-Contrast CT scan
* Presence of active HEENT infection including acute dacryocystitis, with the exception of CRS infection
* Febrile illness within 2 weeks of procedure and/or active pus from nose
* Any sign of active ophthalmic disease, infection, or inflammation including the presence of severe ocular surface inflammatory disease as determined by ophthalmic and physical exam, which could be exacerbated by the presence of the device
* Best Corrected Visual Acuity (BCVA) worse than 20/50
* Dry Eye disease defined by the following:
* Abnormal Tear Breakup Test (TBUT) (< 5 seconds) in either eye and
* Corneal staining showing superficial punctate keratopathy of Grade 1 or higher in either eye at Screening Visit
* Use of topical or systemic prescription ocular medications, except rewetting drops for contact lens-related discomfort, for the eye to treat an active ophthalmic disease at or within 14 days of screening and through procedure
* Underlying medical condition that, in the opinion of the Investigator, would place the subject at high risk if IV sedation (MAC or monitored anesthesia care) were used during the procedure
* Excessive ocular and/or adipose tissue that may obscure implanted device visualization and/or placement
* Known allergies to silicone, TobraDex® (Tobramycin and Dexamethasone), procedural medications, and ophthalmic eye drops (required for routine eye exams)
* Documented diagnostic history of Cystic Fibrosis
* Documented history of migraines, cluster headaches, chronic daily headaches or other headaches unrelated to the sinus
* Documented uncontrolled or poorly controlled seasonal or perennial allergies
* Requires any amount of concurrent systemic steroid medication for chronic illness such as auto-immune diseases
* Tobacco, marijuana and/or e-vape inhaler use either currently or during the last 90 days
* Documented history of bleeding disorders, for example, von Willebrand's disease or hemophilia
* Inability to stop thrombolytics or other anti-platelet medication prior to procedure day including but not limited to Coumadin (warfarin) for 5 days, Plavix (clopidogrel) for 3 days, ASA/NSAIDs/fish oil supplements for 10 days, Xarelto® (rivaroxaban) for 24 hours
* For contact lens wearers, inability to go without contact lenses for at least 10 days postoperatively
* Known use of any investigational ocular or sinus drug(s) or devices within 30 days prior to enrollment
* Investigator determination that the potential study subject is unable to comply with study procedures and/or follow-up, or provide informed consent
* Women of childbearing potential who test positive on the study-required urine pregnancy test or who are unwilling to practice a medically acceptable contraception regimen from Screening Visit though Week 12 visit. Women who are documented as postmenopausal for at least 1 year (> 12 months since last menses) or are surgically sterilized do not require testing
* Severe co-morbidity or poor general physical/mental health that, in the opinion of the Investigator, will not allow the subject to be a good study candidate (i.e. other disease processes, mental capacity, cognitive function, substance abuse, shortened life expectancy, vulnerable patient population, high surgical risk)
* Currently involved in another clinical study where that participation may conflict or interfere with the treatment, follow-up or results of this clinical study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Zinreich CT Score | 12 Weeks
  The average change in the Zinreich modified Lund-Mackay scoring of CTs (Zinreich Modified CT) from screening to 12 Weeks

SECONDARY OUTCOMES:
SNOT-22 Score | 12 Weeks
  Intermediate changes from Screening in the Total SNOT-22 will be calculated from screening to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joel Hale, Study Director — Sinopsys Surgical
Locations (6):
- United States (6):
  - Front Range ENT, Greeley, Colorado
  - Ear, Nose & Throat Associates of South Florida, Boca Raton, Florida
  - Kentuckiana Ear, Nose & Throat, PSC, Louisville, Kentucky
  - The Rontal Clinic, Farmington Hills, Michigan
  - Madison ENT, New York, New York
  - EVMS Otolaryngology, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No